CLINICAL TRIAL: NCT07066969
Title: Investigating the Prevalence of Germline Alterations in Actionable Genes in Endometrial Cancer
Brief Title: Prevalence of Germline Alterations in Actionable Genes in Endometrial Cancer
Acronym: GerEC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UID 4914; UID 4914 (Other: Clinical Trial Office - Istituto Europeo di oncologia)
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endometrial Cancer patients with tumoral BRCA (Other): Patients with diagnosis of endometrial cancer
  Interventions: Genetic: Sophia DDM

INTERVENTIONS:
Genetic: Sophia DDM — Germline panel for patients with tumoral BRCA alteration in EC

SUMMARY:
Endometrial cancer (EC) is the most common gynecological cancer in developed countries, with 10200 new cases of EC (5.5% of all cancers) estimated in 2023 and 2500 death for EC estimated in 2022 in Italy.

Recently, the classical clinicopathological risk factors, such as age, FIGO stage, myometrial invasion, tumor grade, lymphovascular space invasion, and lymph node status, have been associated with molecular features for EC risk stratification. The recently introduced molecular classification, based on a very relevant publication of the "Integrated genomic characterization of endometrial carcinoma" by The Cancer Genome Atlas research network in 2013,2 requires the evaluation of three surrogate molecular markers, namely POLE sequencing, p53 immunohistochemical (IHC) evaluation, and mismatch repair (MMR) protein IHC evaluation, in order to reproduce the TCGA model and translate it into clinical practice.

This molecular-based risk stratification provides a more accurate prediction of recurrent or metastatic disease than traditional clinicopathological criteria; however, more molecular knowledge is needed to better understand EC. Recently, the European Institute of Oncology implemented a new molecular panel for somatic evaluation of EC (Sophia DDM). The panel includes 54 genes, including BRCA1 and BRCA2.

DETAILED DESCRIPTION:
Endometrial cancer (EC) is the most common gynecological cancer in developed countries, with 10200 new cases of EC (5.5% of all cancers) estimated in 2023 and 2500 death for EC estimated in 2022 in Italy. Recently, the classical clinicopathological risk factors, such as age, FIGO stage, myometrial invasion, tumor grade, lymphovascular space invasion, and lymph node status, have been associated with molecular features for EC risk stratification. The recently introduced molecular classification, based on a very relevant publication of the "Integrated genomic characterization of endometrial carcinoma" by The Cancer Genome Atlas research network in 2013,2 requires the evaluation of three surrogate molecular markers, namely POLE sequencing, p53 immunohistochemical (IHC) evaluation, and mismatch repair (MMR) protein IHC evaluation, in order to reproduce the TCGA model and translate it into clinical practice. The 4 molecular categories proposed are the following: 1) POLE-mutated, identified by pathogenic variants (PV) in polymerase epsilon exonuclease (POLE) gene; 2) non-specific molecular profile (NSMP); 3) mismatch repair deficient (MMRd)/microsatellite instability; 4) p53 abnormal (p53abn), determined by copy number variations and PV in TP53. Based on the results of these studies, current European guidelines3,4 and 2023 FIGO staging5 integrated the molecular categories to the histological features for EC staging, risk classification, and adjuvant treatment recommendation. Since then, the evaluation of the three molecular surrogates has become more widely used. While p53 and MMR proteins can be evaluated by IHC, POLE has to be evaluated by sequencing.

This molecular-based risk stratification provides a more accurate prediction of recurrent or metastatic disease than traditional clinicopathological criteria; however, more molecular knowledge is needed to better understand EC. Recently, the European Institute of Oncology implemented a new molecular panel for somatic evaluation of EC (Sophia DDM). The panel includes 54 genes, including BRCA1 and BRCA2.

The role of BRCA and other actionable genes alterations in endometrial cancer Several studies have investigated the prevalence of endometrial cancer (EC) in individuals carrying germline BRCA1 and BRCA2 PV, suggesting a potential association between BRCA PV and increased EC risk.6-9 Emerging evidence indicates that germline BRCA PV carriers are at a heightened risk of developing serous EC compared to the general population. For instance, a recent metanalysis reported that women with BRCA PV had a higher observed-to-expected ratio of uterine serous carcinoma (17.97; 95% CI; p<0.001).9 In addition, there is debate about whether BRCA PV carriers have an increased risk of endometrial cancer overall, with studies reporting conflicting results. A systematic review and meta-analysis by Matanes et al.10 showed a slightly increased risk of EC, particularly among BRCA1 carriers. Another meta-analysis by Nahshon et al.9 reported a standardized incidence ratio (SIR) of 2.22 for EC among BRCA mutation carriers. Zakerinasab et al.11 further corroborated these findings, suggesting that BRCA1/2 carriers have approximately a two-fold increased risk of EC.

Despite these findings, comprehensive data on the overall frequency of somatic and germline BRCA PV across all histologic subtypes of EC remain scarce. This gap in knowledge underscores the need for further investigation into the broader role of BRCA genes in EC pathogenesis.

In our study, utilizing the Sophia DDM panel, Tumoral BRCA PV has been detected in 9.7% of EC cases, a frequency significantly higher than previously reported estimates (4.3% according to a recent systematic review by Gasparri et al.12 Notably, in our cohort of unselected EC patients undergoing primary surgery-distinct from previously published cohorts-tumoral BRCA PV were identified in endometrioid EC cases. While previous studies have highlighted the link between BRCA PV and serous EC,6,7,13 our findings suggest a broader role, extending to endometrioid EC. This finding challenges the prevailing assumption that BRCA PV are predominantly associated with serous histology. Intriguingly, the majority of these BRCA-mutated endometrioid EC cases exhibited co-occurring alterations in genes implicated in distinct molecular EC subgroups, such as POLE (ultramutated), mismatch repair genes (MMRd), or TP53 (p53abn).

The frequency of tumor-positive PV in actionable genes, including BRCA1, BRCA2, MSH2, MSH6, PMS2, MLH1, EPCAM, POLE, TP53, PTEN, suggests that germline testing for these genes in patients with EC is critical to identify mutations that can guide personalized treatment plans, inform surveillance strategies for patients and their families, and potentially improve outcomes through early detection and prevention of secondary cancers.

Currently, germline genetic testing data for this cohort are unavailable, limiting our understanding of the association between somatic and germline BRCA PV. This distinction is crucial for assessing hereditary cancer risk and guiding targeted therapeutic strategies. Further studies integrating germline genetic analysis are warranted to clarify the clinical significance of somatic BRCA PV in EC and their potential as biomarkers for prognosis or therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of EC
* tumoral BRCA mutation

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of actionable germline alterations in tBRCA mutated endometrial cancer. | 18 months
  Genomic DNA will be extracted from peripheral blood leukocytes and analyzed with the SOPHiA DDM™ Hereditary Cancer Solution (HCS) v2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Betella, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided